CLINICAL TRIAL: NCT06054490
Title: Self-management and Home Exercises for the Treatment of Masticatory Muscle Pain. A Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional Andres Bello (Other)
Responsible Party: Principal Investigator, Javier Salinas Aguilar, Clinical Professor, Universidad Nacional Andres Bello
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10.17605/OSF.IO/EFBC2
Record Dates: First submitted 2023-09-08; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Myalgia of Mastication Muscle
Keywords: temporomandibular joint disorders; myalgia; self-care; self-management
MeSH Terms: conditions — Temporomandibular Joint Disorders; Myalgia | interventions — Self-Management

STUDY DESIGN:
Intervention Model Description: The patients were contacted by telephone the day before each session appointment to avoid dropouts and to remember to keep an exercise record if applicable. The treatment of the subjects consisted of 5 sessions. (S1) evaluation and diagnosis of recruited subjects; (S2) three days after S1, SM instruction and explanations of the follow-up sessions were given to all subjects, in addition home exercises were instructed and explained to the SM+EX group; (S3) first control and reinforcement of SM (or SM and exercises) at 2 weeks; (S4) second control and reinforcement of SM (or SM and exercises) at 6 weeks; (S5) third control and is encouraged to continue with SM. Referral to a specialist is made if initial symptom remission has not been achieved.
Who Masked: Participant, Outcomes Assessor
Masking Description: In the first session, the operator explained to the study subjects the alternatives, benefits and possible complications of the treatments, it was also indicated that at the time of treatment administration they would not be explained to which group they were assigned to protect the blinding of the treatments. The study of the information was carried out with the necessary precautions to allow masking and blinding of the results obtained, achieving an objective analysis of the results by the outcomes assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-management group (SM group) (Active Comparator): Subjects in this group received a scheme of self-management protocol consisting of verbal and written information on the etiology and prognosis of TMD.
  Interventions: Behavioral: Self-management; Other: Home exercises
- Self-management plus home exercises group (SM+EX group) (Experimental): Subjects in this group received self-management protocol in combination with a home self-exercise routine. Basic exercise therapy includes mobilization, stretching, and muscle strengthening exercises.
  Interventions: Other: Home exercises

INTERVENTIONS:
Behavioral: Self-management — It is based on the premise that cognition, the process of acquiring knowledge and forming beliefs, is a primary determinant of mood and behavior. The therapy uses self-management techniques to identify, correct and prevent behaviors or situations capable of altering the subject's state. In addition, relaxation techniques, sleep hygiene, diet modification, thermotherapy, encouragement to practice social and aerobic activities, and how to prevent risk factors and bad habits.
  Other Names: SF
  Arms: Self-management group (SM group)
Other: Home exercises — It is based on home self-exercise routine. Basic exercise therapy includes mobilization, stretching, and muscle strengthening exercises
  Other Names: EX

SUMMARY:
The objective of this study was to compare the clinical effectiveness of self-management (SM) together with mandibular home exercises (EX) in the treatment of myalgia of the masticatory muscles. A controlled clinical trial was carried out with a total of 48 subjects diagnosed with myalgia according to the diagnostic criteria for temporomandibular disorders (DC/TMD), who were randomized into two groups: treated with SM (SM group) and treated with SM and mandibular home exercises (SM-EX group). The follow-ups were carried out at 2, 6 and 10 weeks, where the following were evaluated: pain in the masticatory muscles, range of mandibular movement and mandibular functional limitation.

DETAILED DESCRIPTION:
Materials and method. This randomized controlled clinical trial was conducted between January 2016 and June 2016 at the Andres Bello University Dental Clinic (Viña del Mar, Chile). Study subjects were recruited from the universe of patients seeking treatment for jaw pain at the School of Dentistry. All subjects were informed about the study by their operator and gave their written consent before beginning the study. The protocol, design, and implementation were approved by the Scientific Ethics Committee of the Faculty of Dentistry of the Andres Bello University, Viña del Mar, Chile (Folio No. 056, year 2016). Which was in accordance with the latest version of the Declaration of Helsinki of the World Medical Association (Declaration of the World Medical Association of Helsinki, 2013).

Sample's size calculation. An error percentage of 7% was calculated according to a confidence level of 91%, considering a prevalence of chewing muscle pain of 9% and an expected loss of 1.08% based on the losses obtained in the study carried out by Kalamir. et al. in 2012 (Kalamir et al., 2012). The minimum number of participants required for each group was 25 patients (50 patients in total).

Randomization and interventions. After meeting the inclusion and exclusion criteria, subjects were randomly assigned to two groups using a computer generated sequence "random list" developed by random.org.

Evaluation methods. The initial evaluation, to determine the degree of involvement of axis I, was carried out following the symptom questionnaire and clinical examination guidelines according to the DC/TMD protocol. Additionally, the questionnaire for the chronic pain grade scale (GCPS v2.0) and the functional limitation scale (JFLS-20) of axis II of the DC/TMD protocol were applied. In turn, an intraoral clinical examination was performed to rule out pain of dental origin.

Statistic analysis. Demographic characteristics of the sample were reported descriptively. Data were analyzed using Wilcoxon signed-rank test for comparisons between periods (initial evaluation, and weeks 2, 6, and 10) and Wilcoxon rank-sum test for comparison between groups of the variables MMP, MRM, JFLS-20. Qualitative evaluation of adherence to self-management was analyzed using Fisher exact test. Qualitative evaluation of adherence to home exercises was descriptively reported. The level of significance was established at p=0.05. All statistical analysis was performed using R-Crain 3.01 software.

ELIGIBILITY:
Inclusion Criteria:

* "Age between 18 and 40 years", "Presence of myalgia of the masticatory muscles according to DC / TMD diagnostic criteria."

Exclusion Criteria:

* "Painful joint TMD"; "history of treatment for TMD"; "recent history of facial or cervical trauma"; "ongoing orthodontic treatment"; "Tooth mobility secondary to periodontal disease"; "Subjects with loss of more than two teeth other than third molars and / or premolars due to orthodontic indication"; "subjects with systemic musculoskeletal diseases or who are under analgesic treatment"; "Subjects with a diagnosed intellectual disability who cannot express their will to participate in scientific research as established by law 20.584 of Chile."

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Masticatory muscle pain (MMP) | It was applied in the initial evaluation, week 2, 6 and 10
  Pain intensity was measured using a verbal numeric scale (VNS); subjects were asked to verbally rate the perceived intensity using a numerical rating scale where "0" corresponded to "no pain" and "10" corresponded to "extremely strong pain"

SECONDARY OUTCOMES:
Mandibular range of motion (MRM) | It was applied in the initial evaluation, week 2, 6 and 10
  Maximum mouth opening in an autonomous and comfortable way, that is, without feeling pain and not assisted by the operator, measured in millimeters from incisal edge to incisal edge of anterior teeth, compensating for overbite
Jaw functional limitation (JFLS-20) | It was applied in the initial evaluation and week 10
  Scale in charge of globally assessing masticatory limitation, vertical mobility limitation, verbal and non-verbal communication limitation, included within a 20-item instrument thanks to the survey of mandibular functional limitation of the DC / TMD. This scale has a score of 0 to 10, with 10 being a severe limitation
Qualitative evaluation of adherence to self-management | It was applied in the initial evaluation, week 2, 6 and 10
  Qualitative evaluation of subjects' adherence to a self-care protocol scheme that was categorized as "good" (⅔ of the time), "moderate" (between ⅔ and ⅓ of the time), and "deficient" (less than ⅓ of the time). Recorded in a "behavior and self-care log per session"
Qualitative evaluation of adherence to home exercises | It was applied only to the SM+EX group in weeks 2, 6, and 10
  Qualitative evaluation of subjects' adherence to a routine self-exercise therapy at home, as recorded in a "patient diary" that was categorized as "good" (⅔ of the time), "moderate" (between ⅔ and ⅓ of the time) and "deficient" (less than ⅓ of the time).

CONTACTS AND LOCATIONS:
Overall Officials: Diego De Nordenfycht, Principal Investigator — Universidad Nacional Andres Bello

IPD SHARING:
Plan to Share IPD: Yes
All the collected IPD, study protocol, statistical analysis plan, informed consent form and a clinical study report will be shared, including results, discussion and bibliography studied.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: One-year database availability period, starting August 28, 2023
Access Criteria: Database will be shared in Open Security Foundation (OSF), a non-profit public organization founded as a support organization for open source security projects.
URL: https://osf.io/efbc2/

REFERENCES:
- [Background] Kalamir A, Bonello R, Graham P, Vitiello AL, Pollard H. Intraoral myofascial therapy for chronic myogenous temporomandibular disorder: a randomized controlled trial. J Manipulative Physiol Ther. 2012 Jan;35(1):26-37. doi: 10.1016/j.jmpt.2011.09.004. Epub 2011 Nov 10. PMID 22079052
- See also: Description The DC/TMD is intended for use in both clinical settings and applied research settings. — https://ubwp.buffalo.edu/rdc-tmdinternational/tmd-assessmentdiagnosis/dc-tmd/
- Available data/document: Study Protocol: 10.17605/OSF.IO/EFBC2 — https://osf.io/efbc2/ — Supporting information for this study is available in the open science framework (OSF): the data set of individual participants, study protocol, statistical analysis plan, and informed consent form